CLINICAL TRIAL: NCT04644900
Title: Effect of Chewing Gum and Mouthwash Before Operation on Sore Throat After General Anesthesia With a Laryngeal Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Director, Principal Investigator, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Na Chen
Record Dates: First submitted 2020-11-22; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Sore Throat
Keywords: sore throat, Laryngeal Mask , Chewing Gum , Mouthwash
MeSH Terms: conditions — Pharyngitis | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Mouthwash group (Active Comparator): Patients in the mouthwash group received 15 ml of honeysuckle antibacterial mouthwash and vomited it out after 2 minutes
  Interventions: Other: Mouthwash
- the gum group (Active Comparator): patients in group gum chewed one piece of herbal sugar-free gum for 2 minutes and then spat it out.
  Interventions: Other: chewed mint gum

INTERVENTIONS:
Other: chewed mint gum — In the preoperative waiting area before transferring to the operating room,patients in group G chewed mint gum for 2 minutes and then spit it out.
  Arms: the gum group
Other: Mouthwash — Patients in the mouthwash group took 15 ml honeysuckle antibacterial mouthwash in their mouths, and vomited them out after 2 minutes
  Arms: the Mouthwash group

SUMMARY:
Postoperative sore throat (POST) is an important problem after general anaesthesia. We assessed whether chewing gum preoperatively or mouthwash can reduce the incidence of POST after general anaesthesia administered via a streamlined liner of the pharyngeal airway (SLIPA).

ELIGIBILITY:
Inclusion Criteria:

American Society of Anaesthesiologists(ASA)class I or II 20~65 years body mass index(BMI)scores<30 undergoing elective hysteroscopic surgery

Exclusion Criteria:

chronic laryngitis chronic bronchitis asthma gastroesophageal reflux allergies to study drugs recent use of non-steroidal anti-inflammatory drugs(NSAIDS) a history of upper respiratory tract infection in the past one week Mallampati grade>2 a history of steroid therapy.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of POST scores>3 | within 24 hours after surgery.
  POST was evaluated by the Numerical Rating Scale(NRS),which ranges from 0 to 10 points,with 0 indicating completely painless,1~3 indicating mild discomfort,4~6 indicating moderate pain,and 7~10 indicating severe pain .

SECONDARY OUTCOMES:
the POST scores | 2 hours,6 hours and 24 hours after surgery.
  POST was evaluated by the Numerical Rating Scale(NRS),which ranges from 0 to 10 points,with 0 indicating completely painless,1~3 indicating mild discomfort,4~6 indicating moderate pain,and 7~10 indicating severe pain .

OTHER OUTCOMES:
subgroup analysis with patient subdivided based on whether the laryngeal mask had blood on it. | Immediately after removal of laryngeal mask
  blood stain

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of The Obstetrics and Gynecology Hospital, Fudan University,, Shanghai, China